CLINICAL TRIAL: NCT04909138
Title: Intermittent Dosing of Dorsal Root Ganglion Stimulation as an Alternate Paradigm to Continuous Low-Frequency Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Sandeep Amin, MD, Principal Investigator- Anesthesia Department (Provider), Rush University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 21051403
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: CRPS (Complex Regional Pain Syndromes); Radiculopathy; Peripheral Neuropathy
Keywords: Chronic Pain; Dorsal Root Ganglion Stimulation
MeSH Terms: conditions — Complex Regional Pain Syndromes; Radiculopathy; Peripheral Nervous System Diseases; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Patients will be prospectively randomized to one of two stimulation paradigms both of which involve intermittent dosing at 30 seconds ON and 90 seconds OFF. Group 1 will have their frequency set at 20 Hz with amplitude set just below perception. Group 2 will have their frequency set at 5 Hz with amplitude set just below perception. This study will be performed in a crossover fashion with a washout period, meaning patients will receive one of the stimulation parameters at baseline, return to their pre-study stimulation settings at the 12-week time period and receive the alternate stimulation dosing regimen at the 13-week time period.
Who Masked: Participant
Masking Description: Participants will not know to which treatment they are randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- DRG stimulation therapy at 20 Hz and 30 seconds ON, 90 seconds OFF (Active Comparator): DRG stimulation therapy at 20 Hz (30 seconds ON, 90 seconds OFF)
  Interventions: Device: DRG stimulation 20 Hz 30/90
- DRG stimulation therapy at 5 Hz and 30 seconds ON, 90 seconds OFF (Active Comparator): DRG stimulation therapy at 5 Hz (30 seconds ON, 90 seconds OFF)
  Interventions: Device: DRG stimulation 5 Hz 30/90

INTERVENTIONS:
Device: DRG stimulation 20 Hz 30/90 — Stimulation delivered at 20 Hz and 30 seconds ON, 90 seconds OFF
  Arms: DRG stimulation therapy at 20 Hz and 30 seconds ON, 90 seconds OFF
Device: DRG stimulation 5 Hz 30/90 — Stimulation delivered at 5 Hz and 30 seconds ON, 90 seconds OFF
  Arms: DRG stimulation therapy at 5 Hz and 30 seconds ON, 90 seconds OFF

SUMMARY:
This study seeks to evaluate the use of intermittent dosing as an alternative paradigm for patients with DRG stimulation in place for at least 1 year and minimum 50% pain relief in the targeted area.

Patients will be prospectively randomized to one of two stimulation paradigms both of which involve intermittent dosing at 30 seconds ON and 90 seconds OFF. Group 1 will have their frequency set at 20 Hz with amplitude levels adjusted in order to remain in the therapeutic window (subthreshold stimulation). Group 2 will have their frequency set at 5 Hz with amplitude levels adjusted in order to remain in the therapeutic window (subthreshold stimulation) This study will be performed in a crossover fashion, meaning patients will be changed to the alternate dosing regimen at the 13-week time period.

Patients will be seen and evaluated prior to randomization and reprogramming, and thereafter evaluated at 4, 8, and 12-weeks. At the 12-week time period, patients will begin a 1-week washout period of continuous stimulation. At the 13-week time period, patients will be evaluated, crossed over to the other study arm and thereafter evaluated at 17, 21, and 25-weeks.

DETAILED DESCRIPTION:
Dorsal Root Ganglion (DRG) is a novel target of neuromodulation that's use has grown as a proven effective treatment in chronic painful conditions. Studies examining tonic, paresthesia-based dorsal column stimulation have demonstrated plateauing or diminishing effects after extended time periods. Although not yet studied in DRG stimulation due to its relative infancy, the possibility of decreased pain relief over time very much exists. In order to mitigate the potential for waning pain relief over time, other paradigms of stimulation within the framework of DRG therapy must be evaluated.

Intermittent dosing (ID) refers to the cycling of stimulation, in which there is a designated time period of stimulation being active (ON) and inactive (OFF). Previous studies have demonstrated the safe and effective use of intermittent dosing using spinal cord stimulation (SCS).9,10 In 2020, Deer et al. reported the efficacy of intermittent dosing of Burst stimulation with settings ranging from 30 seconds ON and 90 seconds OFF, to 30 seconds ON and 360 seconds OFF in SCS.10 However, no studies have examined the use of ID in DRG stimulation. Furthermore, a pre-clinical study by Chao et al. 2020 showed that DRG field stimulation delivered at 20 Hz continuously abated transmission of action potentials in most C-type fibers and 50% of Aδ fibers. Conversely, DRG field stimulation delivered at 5 Hz consistently evoked action potentials in Aβ, Aδ, and C type fibers, suggesting that this frequency may have greater potential to mitigate pain11. Nevertheless, translation of these results to clinical practice have yet to be studied.

Patients with chronic pain secondary to CRPS or other chronic neuropathic who have responded to DRG stimulation originally and have undergone permanent DRG stimulator implantation delivered by the Abbott PROCLAIM Dorsal Root Ganglion Neurostimulator System, have had the system in place for at least 1 year, utilizing continuous tonic therapy, reporting minimum 50% pain relief in the targeted area, will be randomized to 1 of 2 study arms, in a single-blinded, 1:1 fashion:

1. High ID Arm: DRG stimulation therapy at 20 Hz frequency for 30 seconds ON, 90 seconds OFF
2. Low ID Arm: DRG stimulation therapy at 5 Hz frequency for 30 seconds ON, 90 seconds OFF

Based on the stimulation frequency each patient receives the stimulation amplitude will be adjusted accordingly to remain in the therapeutic dosing window for each patient.

Patients will be seen and evaluated prior to randomization and reprogramming, and thereafter evaluated at 4, 8, and 12-weeks. At the 12-week time period, patients will begin a 1-week washout period of continuous stimulation at their pre-study stimulation settings. At the 13-week time period, patients will be evaluated, crossed over to the other study arm and thereafter evaluated at 17, 21, and 25-weeks.

As our primary endpoint, we hypothesize that intermittent dosing with either 20 Hz frequency (high) or 5 Hz frequency (low) ID will provide superior pain relief as measured by VAS scores when compared to continuous DRG stimulation therapy in this patient population. Other endpoints include: EQ-5D scores of wellbeing; PROMIS score for physical function, pain interference, sleep disturbance, and emotional distress; chronic pain acceptance questionnaire 8 (CPAQ-8), patient satisfaction scores, and patient global impression of change.

After evaluation, all eligible and consented subjects will be randomized into one of two treatment groups. Randomization will be performed using a computer-generated random sequence generator with equal selection probabilities to all groups. Subjects will be blinded to their randomization.

After randomization, each consented subject will present to clinic at which time will first be seen by a team of investigators, sub-investigators, and/or study staff. Patients will be sent for x-ray at initial presentation to evaluate for real-time DRG lead position. Patients will be excluded from study if there is significant migration, at the discretion of clinician. Patients will have had at least one prior attempted reprogramming in standard fashion (increasing amplitude firing in tonic stimulation to document stimulation is targeting dermatome of initial placement) before enrollment in this study. Otherwise, after evaluation and collection of baseline data, a clinical specialist for the Abbott PROCLAIM Dorsal Root Ganglion Neurostimulator System will program the subject's DRG system according to the treatment group to which they have been randomized, under direct physician supervision and with use of the radiographic films.

Patient will be subsequently evaluated at 4, 8 and 12 weeks. At the 12-week time interval, the patient will begin a 1-week washout period of continuous stimulation. At the 13-week time interval, the patient will be crossed over to the alternative study arm. Thereafter, they will be evaluated again at the 17-week, 21-week, and 25-week time interval. At each interval, the patient will be evaluated by a team of investigators, sub-investigators, and/or study staff to administer questionnaires and collect data.

Patient specific data to be collected prior to first allocated dosing stimulation will include:

* Age
* Height
* Weight
* BMI
* Gender
* Primary diagnosis
* Current daily morphine milligram equivalent usage

Data to be collected at baseline and at 12, 13 and 25 weeks of stimulation only:

* Patient Health Questionnaire (PHQ-8)
* PROMIS Health questionnaires

  * Global Health 10 item questionnaire
  * Physical Function 8b questionnaire
  * Emotional Distress-8a Anxiety questionnaire
  * Sleep Disturbance 4a questionnaire
  * Fatigue 8 item questionnaire
* CPAQ-8 score (Chronic Pain Acceptance Questionnaire 8)
* Patient Global Impression of Change (see fig. 2)
* Patient Satisfaction Score (7-point Likert-type scale; see fig. 2)

Data to be collected at each study visit:

* NRS pain scores (22-point scale, 0-10 in 0.5 increments)
* Current dorsal root ganglion stimulation parameters (i.e. mode of stimulation-continuous vs. ID, frequency, amplitude, pulse width)
* Average charging frequency over last week

Risks & Benefits:

As with all clinical research, there exists a potential for loss of confidentiality. Measure to protect the confidentiality of study participants will be implemented as described in the Data Collection & Management Section Below.

Further loss of therapeutic pain relief is another potential risk that could occur following reprogramming to ID parameters. If at any point a subject reports diminishing pain relief and wishes to return to baseline mode of stimulation, they will be allowed to do so and considered a study failure. Patients would be encouraged to proceed with randomization process and if pain relief diminished, would be allowed to return to whichever desired mode of stimulation.

Subjects may experience benefit in the form of pain relief and improved functionality following reprogramming to ID parameters. However, if the patient chooses to no longer participate in the study, they may still receive treatment from the treating physician, which may include the ID parameters, administered separately, being investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 99
* 1-year or more use of continuous DRG therapy as delivered a permanently implanted Abbott PROCLAIM XR Dorsal Root Ganglion Neurostimulator System for chronic back and/or leg pain
* Endorse at least 50% pain relief in the targeted area over the last year
* Must have been seen for routine follow-up within last 4 months
* Must have been reprogrammed in standard fashion at least once prior to randomization
* Willing and able to complete protocol requirements, including:

  * Complete health questionnaires and pain scales as specified in the protocol
  * Sign the study-specific informed consent form
  * Complete follow-ups at the designated time periods

Exclusion Criteria:

* Significant lead migration, as determined by clinician
* Other concurrent neuromodulation system in place
* Corticosteroid injection in previous 30 days prior to enrollment
* Intermittent dosing and/or failure within last 6m
* Changing or unstable pain medications within 30 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
NRS pain scores | Up to 6 months
  Subject's Numeric Rating Scale (NRS) score for pain being treated by DRG simulation for up to 3 months of designated treatment on a 22 point scale from 0-10 in 0.5 increments with 0 being no pain to 10 being the worse imaginable pain.

SECONDARY OUTCOMES:
Patient Satisfaction with Treatment Score | Up to 6 months
  At each study visit, subjects will rate their satisfaction with their current DRG stimulation therapy over the last 3 days on a scale from completely satisfied to completely dissatisfied as either:
  Completely satisfied (best outcome), Very satisfied, Slightly Satisfied, Neither satisfied nor dissatisfied, Slightly dissatisfied, Very dissatisfied, Completely dissatisfied (worse outcome)
CPAQ-8 | Up to 6 months
  At each study visit, subjects will complete the Chronic Pain Acceptance Questionnaire (CPAQ-8) which asks subjects to rate the truth of different statements about their chronic pain (i.e. I live a full life even though I have chronic pain) as either:
  Never true (0), Very rarely true (1), Seldom true (2), Sometimes true (3), Often true (4), Almost always true (5), Always true (6)
Current mode of stimulation | Up to 6 months
  DRG settings as either Burst stimulation at 30 seconds ON/90 seconds OFF, or 30 seconds ON/360 seconds OFF
Stimulator settings- frequency | Up to 6 months
  Subject's current DRG stimulator setting frequency in hertz (Hz)
Stimulator settings- amplitude | Up to 6 months
  Subject's current DRG stimulator setting amplitude in milliamps (mA)
Stimulator settings- pulse width | Up to 6 months
  Subject's current DRG stimulator setting pulse width in microseconds (μs)
Charging frequency of DRG stimulator | Up to 6 months
  Average charging frequency over the last week of patient's DRG stimulator in hours/minutes.
PROMIS- Fatigue 8 questionnaire | Up to 6 months
  Fatigue 8 questionnaire outcome at up to 3 months on designated treatment. Subjects will rate statements pertaining to feelings of fatigue (i.e. I feel fatigue...) as not at all (1), a little bit (2), somewhat (3), quite a bit (4), or very much (5).
  Subjects will also rate statements pertaining to frequency of fatigue (i.e. How often did you have push yourself to get things done because of your fatigue) as either never (1), rarely (2), sometimes (3), often (4), or always (5).
PROMIS- Sleep Disturbance 4a questionnaire | Up to 6 months
  Sleep Disturbance 4a questionnaire outcome at up to 3 months on designated treatment. Subjects will rate statements pertaining to quality of sleep (i.e. My sleep was refreshing) as either very much (1), quite a bit (2), somewhat (3), a little bit (4), or not at all (5).
  They will also rate their sleep quality as very poor (5), poor (4), fair (3), good (2), or very good (1).
PROMIS- Emotional Distress- 8a Anxiety questionnaire | Up to 6 months
  Emotional Distress- 8a Anxiety questionnaire outcome at up to 3 months on designated treatment. Subjects will rate statements pertaining to feelings of anxiety (i.e. I felt fearful) as either never (1), rarely (2), sometimes (3), often (4), or always (5).
PROMIS- Physical Function 8b questionnaire | Up to 6 months
  Physical Function 8b questionnaire outcome at up to 3 months on designated treatment. Subjects will rate statements pertaining to ability to do physical tasks (i.e. Are you able to run errands and shop) as either unable to do (1), with much difficulty (2), with some difficulty(3), with a little difficulty (4), or without any difficulty (5).
  They will also rate statements pertaining to any health limitations on physical functions (i.e. Does your health now limit you in lifting or carrying groceries) as not at all (5), very little (4), somewhat (3), quite a lot (2), or cannot do (1).
PROMIS- Pain Interference 6b questionnaire | Up to 6 months
  Pain Interference 6b questionnaire outcome at up to 3 months on designated treatment. Subjects will rate statements pertaining the extent that pain interferes with their life (i.e. How much did pain interfere with your enjoyment of life) as either not at all (1), a little bit (2), somewhat (3), quite a bit (4), or very much (5).
  They will answer how much pain kept them from socializing with others in the past 7 days as either never (5), rarely (4), sometimes (3), often (2), or always (1).
PROMIS- Global Health 10 item questionnaire | Up to 6 months
  Global Health 10 item questionnaire outcome at up to 3 months on designated treatment. Subjects will rate statements pertaining to their overall health (i.e. In general, would you say your quality of life is) as either poor (1), fair(2), good (3), very good (4), or excellent (5).
PHQ-8 | Up to 6 months
  At each study visit, subjects will complete the Patient Health Questionnaire (PHQ-8) which asks subjects to rate over the past 2 weeks how often they feel a particular emotion (i.e. feeling tired or having little energy) as either
  Not at all, Several days, More than half the days, Nearly every day
  If any problems were checked off, subjects will rate how difficult these problems made it to do work, take care of things at home, or get along with others as either:
  Not difficult at all, Somewhat difficult, Very difficult, Extremely difficult
Patient Global Impression of Change | Up to 6 months
  At each study visit, subjects will be asked to rate their progress with the current spinal cord stimulator therapy over the last 3 days compared to their paresthesia DRG therapy as either:
  Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse

CONTACTS AND LOCATIONS:
Overall Officials: Robert McCarthy, PharmD, Study Director — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Available upon reasonable request from principal investigator.

REFERENCES:
- [Background] Kapural L, Yu C, Doust MW, Gliner BE, Vallejo R, Sitzman BT, Amirdelfan K, Morgan DM, Brown LL, Yearwood TL, Bundschu R, Burton AW, Yang T, Benyamin R, Burgher AH. Novel 10-kHz High-frequency Therapy (HF10 Therapy) Is Superior to Traditional Low-frequency Spinal Cord Stimulation for the Treatment of Chronic Back and Leg Pain: The SENZA-RCT Randomized Controlled Trial. Anesthesiology. 2015 Oct;123(4):851-60. doi: 10.1097/ALN.0000000000000774. PMID 26218762
- [Background] Miller JP, Eldabe S, Buchser E, Johanek LM, Guan Y, Linderoth B. Parameters of Spinal Cord Stimulation and Their Role in Electrical Charge Delivery: A Review. Neuromodulation. 2016 Jun;19(4):373-84. doi: 10.1111/ner.12438. Epub 2016 May 6. PMID 27150431
- [Background] Deer T, Slavin KV, Amirdelfan K, North RB, Burton AW, Yearwood TL, Tavel E, Staats P, Falowski S, Pope J, Justiz R, Fabi AY, Taghva A, Paicius R, Houden T, Wilson D. Success Using Neuromodulation With BURST (SUNBURST) Study: Results From a Prospective, Randomized Controlled Trial Using a Novel Burst Waveform. Neuromodulation. 2018 Jan;21(1):56-66. doi: 10.1111/ner.12698. Epub 2017 Sep 29. PMID 28961366
- [Background] Alo KM, Redko V, Charnov J. Four Year Follow-up of Dual Electrode Spinal Cord Stimulation for Chronic Pain. Neuromodulation. 2002 Apr;5(2):79-88. doi: 10.1046/j.1525-1403.2002.02017.x. PMID 22151846
- [Background] Turner JA, Loeser JD, Deyo RA, Sanders SB. Spinal cord stimulation for patients with failed back surgery syndrome or complex regional pain syndrome: a systematic review of effectiveness and complications. Pain. 2004 Mar;108(1-2):137-47. doi: 10.1016/j.pain.2003.12.016. PMID 15109517
- [Background] Hayek SM, Veizi E, Hanes M. Treatment-Limiting Complications of Percutaneous Spinal Cord Stimulator Implants: A Review of Eight Years of Experience From an Academic Center Database. Neuromodulation. 2015 Oct;18(7):603-8; discussion 608-9. doi: 10.1111/ner.12312. Epub 2015 Jun 5. PMID 26053499
- [Background] Pope JE, Deer TR, Falowski S, Provenzano D, Hanes M, Hayek SM, Amrani J, Carlson J, Skaribas I, Parchuri K, McRoberts WP, Bolash R, Haider N, Hamza M, Amirdelfan K, Graham S, Hunter C, Lee E, Li S, Yang M, Campos L, Costandi S, Levy R, Mekhail N. Multicenter Retrospective Study of Neurostimulation With Exit of Therapy by Explant. Neuromodulation. 2017 Aug;20(6):543-552. doi: 10.1111/ner.12634. Epub 2017 Jul 17. PMID 28714533
- [Background] Van Buyten JP, Wille F, Smet I, Wensing C, Breel J, Karst E, Devos M, Poggel-Kramer K, Vesper J. Therapy-Related Explants After Spinal Cord Stimulation: Results of an International Retrospective Chart Review Study. Neuromodulation. 2017 Oct;20(7):642-649. doi: 10.1111/ner.12642. Epub 2017 Aug 18. PMID 28834092
- [Background] Vesper J, Slotty P, Schu S, Poeggel-Kraemer K, Littges H, Van Looy P, Agnesi F, Venkatesan L, Van Havenbergh T. Burst SCS Microdosing Is as Efficacious as Standard Burst SCS in Treating Chronic Back and Leg Pain: Results From a Randomized Controlled Trial. Neuromodulation. 2019 Feb;22(2):190-193. doi: 10.1111/ner.12883. Epub 2018 Nov 19. PMID 30456795
- [Background] Deer TR, Patterson DG, Baksh J, Pope JE, Mehta P, Raza A, Agnesi F, Chakravarthy KV. Novel Intermittent Dosing Burst Paradigm in Spinal Cord Stimulation. Neuromodulation. 2021 Apr;24(3):566-573. doi: 10.1111/ner.13143. Epub 2020 Mar 23. PMID 32202044
- [Background] Chao D, Zhang Z, Mecca CM, Hogan QH, Pan B. Analgesic dorsal root ganglionic field stimulation blocks conduction of afferent impulse trains selectively in nociceptive sensory afferents. Pain. 2020 Dec;161(12):2872-2886. doi: 10.1097/j.pain.0000000000001982. PMID 32658148